CLINICAL TRIAL: NCT04975698
Title: Administration of HIV-specific T Cells to HIV+ Patients Receiving High Dose Chemotherapy Followed by Autologous Stem Cell Rescue - Auto -RESIST BMT CTN 1903
Brief Title: HIV Antigen-specific T-cells Targeting Conserved Epitopes (HST-NEETs) BMTCTN1903
Acronym: BMTCTN1903
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Catherine Bollard (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other); Children's National Research Institute (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Primary Investigator, National Heart, Lung, and Blood Institute (NHLBI)
Organization: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN1903; 2U10HL069294-11 (NIH)
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-09

CONDITIONS: HIV Associated Lymphoma
MeSH Terms: conditions — Lymphoma, Primary Effusion | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HST-NEETs (Other): HIV+ Participants that were treated with autologous hematopoietic stem cell transplant.
  Interventions: Biological: HST-NEETs; Biological: Bone Marrow Transplant

INTERVENTIONS:
Biological: HST-NEETs — HST-NEETs are manufactured from an autologous peripheral blood or MNCs via apheresis collection and will be administered as a single intravenous (IV) infusion of 2x10^7/m^2 cells between 3 Days and 7 Days post-ASCT.
Biological: Bone Marrow Transplant — Day 0 is the day of bone marrow transplantation.

SUMMARY:
This is a Phase II multi-center trial single arm trial of autologous transplantation (ASCT) followed by administration of HST-NEETs for treatment of HIV associated lymphoma

DETAILED DESCRIPTION:
Eligible participants will have 100-120 mL of peripheral blood or 80-100 mL of MNCs via apheresis collected and shipped to Children's National Hospital at ambient temperature. The sample will be used to manufacture the HST-NEET product. The autologous peripheral blood stem cell graft suitable for rescue following conditioning will be obtained either before or after the collection of blood to generate HST-NEETs. Pre-transplant conditioning will consist of BEAM; BCNU 300 mg/m^2 on Day -6, Etoposide 100 mg/m^2 BID and Ara-C 100 mg/m2 BID on Days -5, -4, -3 and -2 and Melphalan 140 mg/m2 on Day -1. ASCT on Day 0. If the mobilized graft contains greater than 5.0 x 106 CD34+ cells per kg, any additional cells should be cryopreserved as a "back-up" graft in the event of graft failure related to the HST-NEETs. Participants will receive one dose (2 x 107 cells/m^2 ) of HST-NEETs between Days +3 to +7 based on the clinical condition of the participant. If this window is missed, the HST-NEETs may be administered up to Day +30 post-ASCT. Participants will be followed for at least one year after ASCT.

ELIGIBILITY:
Eligible participants are HIV positive and plan to be treated by high dose chemotherapy followed by an autologous stem cell transplant (ASCT). Participants are a minimum of 15 years of age with Karnofsky performance status greater than or equal to 70% that have primary refractory or recurrent diffuse large B-cell, immunoblastic, plasmablastic, high grade, Burkitt, primary effusion lymphoma, or classical Hodgkin lymphoma. Participants must have chemosensitive disease as demonstrated by complete or partial response to induction or most recent salvage chemotherapy. Participants cannot have had prior autologous, allogeneic HCT, or CART-cell therapy. Participants must initiate conditioning therapy within 3 months of stem cell mobilization or bone marrow harvest. Blood cell mobilization or bone marrow harvest will be carried out per institutional guidelines. Participants may not have HIV refractory to pharmacologic therapy. Patients must not have an uncontrolled infection. Participants must not have received previous cellular therapy

1. Age 15 years old or older at time of enrollment.
2. Receiving antiretroviral therapies (ART) with HIV viral load < 200 copies or below the limit of detection by standard commercial assay. An HIV-1 RNA measurement that is ≥ 200 copies measured by an FDA-approved commercial assay but <500 copies may be allowed if this is followed by an HIV-1 RNA measurement below the limit of detection or if an exception is approved.
3. Diagnosis of refractory or recurrent diffuse large B-cell lymphoma, composite lymphoma with greater than 50% diffuse large B-cell lymphoma, mediastinal B-cell lymphoma, immunoblastic, plasmablastic, Burkitt or high grade B cell lymphoma or classical Hodgkin lymphoma. Participants with aggressive B-cell lymphoma that is transformed from follicular lymphoma are eligible for the study, pending fulfillment of other criteria.
4. Plan to treat participant with high dose chemotherapy and autologous hematopoietic stem cell transplantation (ASCT).
5. All participants must have chemosensitive disease as demonstrated by at least a partial response (as defined by the criteria in Chapter 3) to induction or salvage therapy.
6. Absolute Lymphocyte Count (ALC) greater than or equal to 800/µL. If ALC is less than 800/uL but still above 400/uL patient may be eligible if the HST-NEETs manufacturing blood product is collected via non-mobilized leukapheresis(apheresis).
7. Participants with adequate organ function as measured by:

   1. Cardiac: Participants must have a left ventricular ejection fraction at rest greater than or equal to 40% demonstrated by MUGA or echocardiogram.
   2. Hepatic:

   i. Bilirubin less than or equal to 2.0 mg/dL (except for isolated hyperbilirubinemia attributed to Gilbert syndrome or antiretroviral therapy as specified in Appendix D) and ALT and AST less than or equal to 3x the upper limit of normal. ii. Concomitant Hepatitis: Participants with chronic hepatitis B or C may be enrolled on the trial providing the above criteria are met. In addition, they must not have evidence of active viral replication by PCR, and no clinical or pathologic evidence of irreversible chronic liver disease. c) Renal: Creatinine clearance (calculated creatinine clearance is permitted based on institutional practice) greater than 40 mL/min.

   d) Pulmonary DLCO (corrected for hemoglobin), FEV1, FVC greater than or equal to 45% of predicted.
8. Voluntary written consent or assent obtained prior to enrollment on study with the understanding that consent or assent may be withdrawn by the participant at any time without prejudice to future medical care.

Exclusion Criteria:

1. Karnofsky performance score less than 70%.
2. Participant is known to have an HIV subtype other than B.
3. Participant has documented raltegravir or protease inhibitor resistance.
4. Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia.
5. Uncontrolled bacterial, viral or fungal infection (currently taking medication and with progression or no clinical improvement).
6. Participant has active CNS involvement.
7. Participants with prior malignancies except resected non-melanoma skin cancer or treated cervical carcinoma in situ. Cancer treated with curative intent greater than or equal to 5 years previously will be allowed. Cancer treated with curative intent less than 5 years BMT CLINICAL TRIALS NETWORK HIV T-Cell - Protocol 1903 Version 1.0 Dated February 24, 2021 2-4 Confidential previously may be eligible must be reviewed and approved by the Protocol Officer or Chairs.
8. Female participants that are pregnant as per institutional definition or breastfeeding.
9. Fertile men or women unwilling to use contraceptive techniques from the time of initiation of mobilization until six-months post-transplant.
10. Prior autologous or allogeneic HCT, or prior therapy with chimeric antigen receptor (CAR) T-cells.
11. Participants with evidence of MDS/AML or abnormal cytogenetic analysis indicative of MDS on the pre-transplant bone marrow examination. Pathology report documentation need not be submitted.
12. Steroids greater than 0.5 mg/kg/day prednisone equivalents.
13. Bone marrow involvement by lymphoma at time of workup. Prior history of bone marrow involvement is allowed if cleared prior to ASCT.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To determine 1.) the proportion of participants who can be treated with (HST-NEETs) within 1 week of ASCT in a cooperative multi-institutional setting and 2.) the efficacy of HSTNEETs in reducing the HIV intact proviral | 6 Months
  Feasibility is defined as a participant receiving HST-NEETs within 1 week post-ASCT; Efficacy will be measured by the reduction in intact proviral reservoir.

SECONDARY OUTCOMES:
Progression-free survival | 6 Months and 1 Year
  Participants are considered a failure for this endpoint if they die or if they relapse/progress or receive anti-lymphoma therapy, other than post-transplant consolidative localized radiation (maximum 3 sites) to sites of prior bulk disease pre-transplant (greater than 3cm)
The incidence and severity of acute infusion related toxicities | 1 Year
  Acute infusion related toxicities are defined as toxicities related to the infusion of HST-NEETs that occur within 24 hours of the infusion.
Impact of therapy on the HIV intact proviral reservoir | 1 Year
  Impact on intact proviral reservoir will be assessed using the IPDA at 4-8 weeks prior to transplant and 12 months following ASCT

OTHER OUTCOMES:
Complete Response(CR) and Complete Response + Partial Response(PR) rates | 100 Days
  CR or PR will be assessed according to the LYRIC criteria
Overall survival | 6 months and 1 year
  Overall survival is defined as death from any cause
Time to hematopoietic recovery | 1 Year
  Time to neutrophil recovery will be the first of three consecutive labs of greater than or equal to 500 neutrophils/μL following the expected nadir. Time to platelet engraftment will be the date platelet count is greater than or equal to 20,000/μL for the first of three consecutive labs with no platelet transfusions 7 days prior.
Incidence of infections | 1 Year
  The incidence of viral, fungal and bacterial infections will be tabulated. All Grade 2 and Grade 3 infections will be reported according to the BMT CTN Technical MOP from Day 0 up to 1 year post-transplant. Infections of interest will be captured and described. The incidence rate of infections is defined by the number of infections divided by the total person-time accumulated over the duration of the study.
Non-relapse mortality | 6 Months 1 Year
  Non-Relapse Mortality (NRM) is defined as death occurring in a participant without relapse progression and will be measured at 6 months and at 1 year.
Toxicities | 1 Year
  Toxicities related to the BEAM conditioning regimen and HST-NEETs infusion beyond the 24 hour acute toxicity monitoring period will be defined by using the version 5.0 CTCAE criteria. All grades of toxicity related to HST-NEETs will be collected. Only grade 3 or higher conditioning regimen related toxicities will be collected.
Assessment of plasma DNA in blood (clonal Ig DNA) as a tumor marker | 100 days, 6 months, 1 year
  Blood specimens will be collected prior to the initiation of conditioning, and at Days 100, 6 months and 1 year post-ASCT. The presence of clonal Ig DNA in plasma will be assessed at each of these time points.
Impact of therapy on the HIV intact proviral reservoir | 100 Days
  Impact on intact proviral reservoir assessed using the IPDA Day 100 post-ASCT as compared to baseline at 4-8 weeks prior to transplant.
HIV RNA in plasma | 100 Days, 6 Months, 1 Year
  HIV RNA in plasma will be measured by a sensitive investigational single copy assay (SCA, detection limit 0.38 copy/ml). Blood specimens will be collected, and plasma HIV RNA measured, at study visits corresponding to those associated with IPDA testing: 4-8 weeks prior to transplant, and at Days 100, 6 months and 1 year post-ASCT.
Impact of therapy on the total proviral HIV DNA | 100 days, 6 months, 1 year
  This assay will be measured at study visits corresponding to those associated with IPDA testing: 4-8 weeks prior to transplant, and at Days 100, 6 months and 1 year post-ASCT. This assay will provide information about the proviral reservoir in patients where the IPDA fails due to sequence variation.
HST-NEETs persistence and expansion in vivo | 100 days, 6 months, and 1 year
  Persistence and expansion of HST-NEETs will be measured by frequency of HIV-1 antigen-specific (gag, pol, nef) CD8+ T-cells by ELIspot at baseline and post-infusion at timepoints at Day 100, 6 months, and 1 year post transplant. Change in T cell responses from baseline to post-infusion, measured by frequency of cells secreting IFN-γ by multimer analysis and/or intracellular cytokine staining and/or ELIspot and/or TCR sequencing will be done depending on PBMC cell numbers available and reagent availability.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Devine, MD, MS, Study Chair — National Marrow Donor Program
Locations (11):
- United States (11):
  - City of Hope National Medical Center, Duarte, California
  - Georgetown, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northside, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering (MSKCC), New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol
Time Frame: Within 6 months of official study closure at participating sites
Access Criteria: Available to public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- See also: Blood and Marrow Transplant Clinical Trials Network Website — https://bmtctn.net/

DOCUMENTS (4):
  • Study Protocol (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT04975698/Prot_001.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04975698/SAP_002.pdf
  • Informed Consent Form: Assent to Participate in Research (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04975698/ICF_004.pdf
  • Informed Consent Form: Informed Consent to Participate in Research (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04975698/ICF_003.pdf